CLINICAL TRIAL: NCT03685916
Title: Screening of Phytochemical Rich Ingredients as 'Functional Foods' to Improve Cardiometabolic Health
Acronym: PRIFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/00258
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Control (Other): 50 grams carbohydrate in the form of rice, 200 milliliters of plain water and 20 grams of garden peas.
  Interventions: Other: Control
- Cumin Rice (Experimental): 50 grams carbohydrate in the form of rice with cumin, 200 milliliters of plain water and 20 grams of garden peas.
  Interventions: Other: Cumin Rice
- Cumin Drink (Experimental): 50 grams carbohydrate in the form of rice, 200 milliliters of cumin extract in solution and 20 grams of garden peas.
  Interventions: Other: Cumin Drink
- Cornsilk Rice (Low dose) (Experimental): 50 grams carbohydrate in the form of rice with cornsilk extract (low dose), 200 milliliters of plain water and 20 grams of garden peas.
  Interventions: Other: Cornsilk Rice (Low dose)
- Cornsilk Rice (High dose) (Experimental): 50 grams carbohydrate in the form of rice with cornsilk extract (high dose), 200 milliliters of plain water and 20 grams of garden peas.
  Interventions: Other: Cornsilk Rice (High dose)
- Cornsilk Drink (Low dose) (Experimental): 50 grams carbohydrate in the form of rice, 200 milliliters of cornsilk extract (low dose) in solution and 20 grams of garden peas.
  Interventions: Other: Cornsilk Drink (Low dose)
- Cornsilk Drink (High dose) (Experimental): 50 grams carbohydrate in the form of rice, 200 milliliters of cornsilk extract (high dose) in solution and 20 grams of garden peas.
  Interventions: Other: Cornsilk Drink (High dose)
- Tamarind Rice (Experimental): 50 grams carbohydrate in the form of rice with Tamarind, 200 milliliters of plain water and 20 grams of garden peas.
  Interventions: Other: Tamarind Rice
- Tamarind Drink (Experimental): 50 grams carbohydrate in the form of rice, 200 milliliters of Tamarind extract in solution and 20 grams of garden peas.
  Interventions: Other: Tamarind Drink

INTERVENTIONS:
Other: Control — Plain rice with plain water
  Arms: Control
Other: Cumin Rice — Cumin rice with plain water
  Arms: Cumin Rice
Other: Cumin Drink — Cumin drink with plain rice
  Arms: Cumin Drink
Other: Cornsilk Rice (Low dose) — Low dose cornsilk rice with plain water
  Arms: Cornsilk Rice (Low dose)
Other: Cornsilk Rice (High dose) — High dose cornsilk rice with plain water
  Arms: Cornsilk Rice (High dose)
Other: Cornsilk Drink (Low dose) — Low dose cornsilk drink with plain rice
  Arms: Cornsilk Drink (Low dose)
Other: Cornsilk Drink (High dose) — High dose cornsilk drink with plain rice
  Arms: Cornsilk Drink (High dose)
Other: Tamarind Rice — Tamarind rice with plain water
  Arms: Tamarind Rice
Other: Tamarind Drink — Tamarind drink with plain rice
  Arms: Tamarind Drink

SUMMARY:
To find out whether consumption of different kinds of plant based functional food ingredients, traditionally used in Asia, can improve post-meal response of indicators of heart and metabolic (cardiometabolic) function.

DETAILED DESCRIPTION:
The study will be a non-blinded, randomised crossover trial with each participants testing between 2 to 4 different test ingredients requiring 5 or 9 separate test sessions (depending on how many the participants opt in for) on 9 non-consecutive days. The number of test ingredients that each participant will consume will be determined by the researcher and communicated to the participant. One of the test sessions will be a control session consisting of plain white rice (50 g available carbohydrates), with 20 g green vegetables being consumed with 200 ml of plain water. On the other hand, the test meal ingredients will be added either to the same amount of rice during preparation or will be added to 200 ml of plain water. The participants will be required to finish the meals within 15 minutes of serving. Appropriate food safety guidelines will be adhered to during the preparation and administration of test meals. We will be testing 20 separate food based traditional ingredients at either one or two doses. 20 participants will be recruited for each test food. Assuming that a minimum 2 test ingredients are tested in each participant up to 200 Chinese male participants aged between 21 and 60 years will be recruited from the general public in Singapore with body mass index between18.5 to 25.0 kg/m2, normal blood pressure (<140/90 mmHg), and fasting blood glucose (<7.0 mmol/L). The exclusion criteria are people who smoke, with any metabolic diseases (such as diabetes, hypertension etc), with glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency), with medical conditions and/ or taking medications known to affect glycemia (glucocorticoids, thyroid hormones, thiazide diuretics), intolerances or allergies to any foods, partake in sports at the competitive and/or endurance levels and individual who intentionally restrict food intake. Interested participants will first attend a consent and screening visit following an overnight fast to go over the informed consent procedure and ascertain their suitability to take part in the study. During this visit, the researchers will discuss the study in more detail and go through the participant information sheet and address any queries that the potential participant may have. If participants are willing to proceed, they will then be asked to sign the informed consent form and complete the screening visit forms and questionnaires. If suitable to proceed, they will then undertake the screening visit measurements including height, weight, waist circumference, body impedance and blood pressure measurements. If suitable at this stage, a finger prick blood glucose measurement will be carried out using the HemoCue® device (Helsingborg, Sweden). The visit should last approximately 1.5 hours. During each of the test days, participants will receive test meals in a random order made with up to 4 different food based test ingredients or the control meal (without any test ingredients). Randomisation of test meals will be done using the =RAND() function in Excel. The ingredients will tested in various doses and/or forms of consumption. The participants will arrive at the study centre following an overnight fast. After a 15 minute rest period, they will have a cannula inserted in their arm to obtain blood samples at regular intervals. There will be 9 blood draws in total per test session: Baseline (0 h, before test meal) and 8 blood samples after test meals at 0.25 h, 0.5 h, 0.75 h, 1.0 h, 1.5 h, 2.0 h, 2.5 h and 3.0 h. At each time point, we will collect 3 ml (about half a teaspoon) of blood. Therefore, for each test day, up to 30 ml blood will be taken and for the entire 9 test sessions, around 270 ml of blood will be collected (around 18 tablespoons) or if the participants only opt in for 5 test sessions, they will donate approximately 150 ml of blood (around 10 tablespoons). The blood samples collected at each timepoint will be measured for glucose, insulin and markers related to the intake of the test meal ingredients. At 4 time points (0 h, 1 h, 2 h and 3 h), seated blood pressure measurements will also be undertaken for 3 times, using an automated sphygmomanometer (Omron, Japan) and the average of the final two blood pressure readings will be taken as that given timepoint. Each test day should take no longer than 4 hours to complete. Participants will be asked to refrain from alcohol and exercise the day before each test day. The study will last between 4 and 12 weeks to compete and each test session will be undertaken on non- consecutive days, dependent on the participants' availability. The participants will be asked to continue with their usual lifestyle during their study participation when they are not attending the test sessions.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Male
* Age between 21 to 60 years
* Body Mass Index between 18.5 to 25.0 kg/m2
* Waist circumference ≤ 90cm
* Fasting blood glucose < 7.0mmol/L
* Blood pressure <140mmHg systolic and < 90mmHg diastolic
* Do not partake in sports at the competitive and/or endurance levels and willing to stop any strenuous activity during or within 24 hours of test days

Exclusion Criteria:

* Smoking
* Allergic/intolerant to any of the test foods to be administered, or any of the following common food and ingredients: eggs, fish, milk, peanuts, and tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, etc.
* Anyone with intentional food restrictions
* People with known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Having metabolic or cardiovascular diseases (such as diabetes, hypertension, heart condition, etc), Having any other diseases involving the small intestine or the colon (e.g., irritable bowel syndrome, inflammatory bowel disease, gastric reflux) or having any liver or kidney disorders or any family history of kidney stones.
* Having medical conditions and/or taking medications known to affect glycemia (glucocorticoids, thyroid hormones, thiazide diuretics),
* Taking any prescribed medication or dietary supplements which may interfere with the study measurements
* Excessive alcohol consumption: consuming ≥ 6 alcoholic drinks per week
* Individuals who have donated blood or taken part in other studies within 4 weeks of study participation.
* Have poor veins impeding venous access
* Have history of severe vasovagal syncope (blackouts or near faints) following blood draws
* Have known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* A team member of the study or is an immediate family member (Immediate family defined as a spouse, parent, child, or sibling, whether biological or legally adopted

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male participants
Enrollment: 20 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Glucose | Up to 180 minutes
  Plasma glucose measured by COBAS

SECONDARY OUTCOMES:
Diastolic and Systolic Blood Pressure | Up to 180 minutes
  Diastolic and Systolic Blood pressure measured by automated blood pressure monitor
Insulin | Up to 180 minutes
  Plasma Insulin measured by COBAS

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore